CLINICAL TRIAL: NCT02518373
Title: An Open-label Volunteer Study of the Effect of G17DT on the Elevation of Plasma Gastrin Levels After Therapy With a Proton Pump Inhibitor (Omeperazole) in Patients With Treated Stage II/III Colorectal Cancer
Brief Title: Effect of G17DT in Patients With Stage II/III Colorectal Cancer
Acronym: CC5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC5
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — gastrin immunogen; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G17DT & Omeprazole (Experimental): * A 14-day washout period
  * An Omeprazole Treatment Period 1 (Day -15 to Day -1)
  * A G17DT treatment period (Day 0 to Day 85)
  * An Omeprazole Treatment Period 2 (Day 86 to Day 100)
  Interventions: Biological: G17DT; Drug: Omeprazole

INTERVENTIONS:
Biological: G17DT — G17DT is a therapeutic immunogen, formulated as a white, sterile, semi-viscous, water-in-oil emulsion (30:70 weight for weight). It was manufactured and supplied by Nova Laboratories Ltd., in glass ampoules containing 0.5 mL at a concentration of 1.25 mg/mL, as a single dose to be administered by intramuscular injection.
  Other Names: PAS, Gastrimmune
Drug: Omeprazole — Proton pump inhibitor used in the treatment of dyspepsia, peptic ulcer disease, gastroesophageal reflux disease, laryngopharyngeal reflux, and Zollinger-Ellison syndrome.

SUMMARY:
This Phase 2 study was an open label, single-center 18-week study to compare basal and meal stimulated plasma gastrin levels before and after treatment with 3 intramuscular injections of 250 µg G17DT, with and without the concomitant administration of Omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 70 years, inclusive
* Written informed consent was provided
* Histologically confirmed Stage II/III colorectal cancer after radical surgery
* A minimum of 3 months elapsed since completion of the chemotherapy for subjects who had received adjuvant chemotherapy
* Subject had recovered from any toxic effects of chemotherapy

Exclusion Criteria:

* Had a known local recurrence of colorectal cancer or presence of metastatic colorectal cancer lesions
* Was using an inadequate method of contraception (determined at the discretion of the investigator), only for women of childbearing potential who were sexually active
* Was unable to comply with the protocol
* Was unable to abstain from H2 receptor antagonists, PPIs or anticholinergics medications for 2 weeks
* Required H. pylori eradication therapy during the study
* Had prior vaccination with G17DT or any other product with a similar mechanism of action
* Had a history of gastric or vagus nerve surgery
* Had any clinically significant laboratory abnormalities and medical conditions which were unexplained, or, in the opinion of the investigator, did not allow for safe entry of the subject into the study
* Had contraindications to intramuscular injections (e.g., bleeding disorders or treatment with anticoagulants [except for aspirin])
* Had serious and unstable cardiovascular or respiratory disease, other malignancy or any other condition that would have jeopardized subject safety or confounded the results
* Had a known hypersensitivity to diphtheria toxoid, G17DT, any of its components or any similar compound
* Had any other condition that might have influenced the plasma gastrin level (e.g., achlorhydria, Zollinger-Ellison syndrome)
* Had used of an investigational drug within the previous month
* Had taken treatments that alter the immune response such as radiotherapy, corticosteroids, and antineoplastic drugs (Inhaled corticosteroids were permitted.)
* Had conditions that impaired the immune response (e.g., acquired immune deficiency syndrome)
* Had a history of drug or alcohol abuse within the past year
* Was unable to accept a standard breakfast for dietary reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-04; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Change in plasma gastrin level. | up to Day 100
  Compare basal and meal stimulated plasma gastrin levels before and after treatment with three intramuscular injections of 250 µg G17DT, with and without the concomitant administration of Omeprazole.